CLINICAL TRIAL: NCT00159237
Title: GR Defect in Peripheral Blood Mononuclear Cells in COPD
Status: Withdrawn | Type: Observational
Why Stopped: Lead Research left the Institute
Sponsor: Imperial College London (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5899N00007
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

INTERVENTIONS:
Procedure: blood test

SUMMARY:
T.to investigate a possible mechanism of the glucocorticosteroid receptors (GR) defect in patients with severe COPD by studying the effect of dexamethasone (Dex) on GR- binding, interleukin production (IL-6/IL-8) and MKP-1 expression in peripheral blood mononuclear cells blood (PBMC)

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe (stage III, Gold) to very severe (stage IV, GOLD) COPD or subjects who are healthy smokers or subjects who are non-smokers
* Written informed consent

Exclusion Criteria:

* Current upper respiratory tract infections
* Any significant disease or disorder (e.g. cardiovascular, pulmonary (other than asthma), gastrointestinal, liver, renal, neurological, musculoskeletal, endocrine, metabolic, malignant, psychiatric, major physical impairment) which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or may influence the results of the study, or the subjects ability to participate in the study
* Subjects not considered capable, as judged by the investigator, of following instructions of the study, e.g. because of a history of alcohol or drug abuse or any other reason

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe (stage III, Gold) to very severe (stage IV, GOLD) COPD or subjects who are healthy smokers or subjects who are non-smokers
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2005-02 (Estimated); Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sergei A Kharitonov, MD PhD, Principal Investigator — Imperial College London
Locations (1):
- Section of Airway Disease, Asthma Lab, Imperial College London, Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No